CLINICAL TRIAL: NCT06748365
Title: Role of Ferritin in the Clinical Presentation and Short-Term Prognosis of Diabetic Ketoacidosis
Brief Title: Serum Ferritin and Prognosis of DKA
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Joseph Medhat Sobhy, resident at internal medicine department, Sohag University
Other Study IDs: Soh-Med--24-12-07MS
Record Dates: First submitted 2024-12-18; First posted 2024-12-27 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Ketoacidosis
Keywords: serum Ferritin; Diabetic Ketoacidosis
MeSH Terms: conditions — Diabetic Ketoacidosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
the aim of this study is to: evaluate the association between serum ferritin levels and the clinical presentation and short-term prognosis of patients with DKA. Specifically, the correlation between its level and the severity of DKA at presentation and determine its prognostic value in predicting short-term outcomes.

DETAILED DESCRIPTION:
Ferritin studies and correlation to acute events like stroke or Mi was done before, however some studies have found a correlation with the degree and prognosis of these diseases and others not. However no study was tried on DKA patients before so the investigators are trying to find if Ferritin would have a relation with patients of Dka and could be used as a prognostic tool (for example we found in this study when level is less than "200" patients mostly has good prognosis) this is just an example or (serrum ferritin turned out to be irrelevant to DKA prognosis as patients would have good prognosis despite number value) and this will be in selected patients according to criteria to exclude any chronic condition in the investigators hospital care units.

ELIGIBILITY:
Inclusion Criteria:

-

All patients with DKA :

1. Adult Aged 18 years old or older .
2. Type 1 DM , type 2 DM
3. Diagnosis of DKA based on the American Diabetes Association criteria: blood glucose >250 mg/dL, arterial pH <7.3, serum bicarbonate <18 mEq/L,

Exclusion Criteria:

1. Patients age less than 18 years old
2. Iron deficiency anemia and iron overload
3. Chronic Inflammatory Diseases: Conditions such as rheumatoid arthritis, systemic lupus erythematosus, and inflammatory bowel disease
4. Acute and chronic infections, including bacterial, viral, and fungal infections
5. Pt presented with other acute complication (MI,stroke)
6. CKD patients
7. Patients with chronic liver diseases
8. Patients with malignancy
9. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with DKA admitted to the emergency department or intensive care units of Sohag university Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
evaluate the association between serum ferritin levels and the clinical presentation and short-term prognosis of patients with DKA. Specifically, the correlation between its level and the severity of DKA at presentation and determine its prognostic value | Through the study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospitals, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided